CLINICAL TRIAL: NCT03892304
Title: Gynecological Health of Adult Women With Cystic Fibrosis: Positive Impact of the Implementation of an On-site Gynecological Consultation
Brief Title: Gynecological Health Improvement of Adult Women With Cystic Fibrosis
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0530
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult women with Cystic Fibrosis: Cohort of 164 women diagnosed with Cystic Fibrosis (CF) who were patients at the Cystic Fibrosis Adult Referral Centre in Lyon, France in 2017 (compared to 155 in 2014). Women attending the CF adult centre in 2017 were asked to complete a written questionnaire.
  Interventions: Other: Self-report written questionnaire

INTERVENTIONS:
Other: Self-report written questionnaire — Patient questionnaire filled-out in presence of clinical nurse. Gynecological options and contraceptive choices were recorded. Close-ended questions used ("yes/no"): contraception use; contraceptive pill use; contraceptive implant; intrauterine device; tubal sterilization; mechanical contraception; other type of contraception use; previous term delivery; gynecological follow-up; previous Pap smear. If "Yes" was noted, more details were requested (contraception name, delivery date, gynecological follow-up frequency, last Pap smear date).
  Other gynecological history and management data not included in the 2014 questionnaire: age at first menstruation, menstrual cycle regularity without hormonal contraception, age at menopause, previous human papilloma virus vaccination, recurrent vulvovaginal candidiasis, urinary incontinence, fertility/infertility data, and infertility treatment with assisted reproductive technologies. Results were compared with those obtained in 2014 (121 women).

SUMMARY:
Following the results of the research team's cross-sectional study conducted in 2014 describing insufficient gynecological care, the research team implemented an on-site gynecological consultation in the adult Cystic Fibrosis (CF) centre in 2015. The study aimed to compare the results of two surveys conducted successively in 2014 and in 2017 on a cohort of women with CF attending the Lyon CF adult referral centre. All the women attending the adult CF center in 2017 were asked to complete the same self-report written questionnaire that was completed in 2014 about their contraceptive choices, gynecological follow-up and cervical screening. Questions concerning gynecological comorbidities were added to the 2017 questionnaire.

This current study aimed to evaluate the impact of the implementation of an on-site gynecological consultation on gynecological health of women with CF, as measured through 3 indicators: the proportion of women with regular gynecological follow-up, cervical screening coverage, and contraceptive coverage. The identification of specific gynecological comorbidities was the other objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* women with cystic fibrosis
* subjects followed by the Cystic Fibrosis Adult Referral Centre in Lyon, France in 2017

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women with Cystic Fibrosis
Study Population: Adult women at least 18 years old diagnosed with Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of women with regular gynecological follow-up | 2014 - 2017
  Comparison of the proportion of patients with a regular gynecological follow-up (at least yearly) between 2014 and 2017.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rousset-Jablonski, MD, Principal Investigator — Hospices Civils de Lyon, Cystic Fibrosis Adult Referral Centre, Department of Internal Medicine, Centre Hospitalier Lyon Sud